CLINICAL TRIAL: NCT06997432
Title: Study of the Clinical and Immunological Implications of Maintaining in the Diet the Maximum Tolerated Dose Identified in a Controlled Food Exposure Test According to the Sensitization Profile to LTPs
Brief Title: Endophenotyping for Plant-based Food Allergy Diagnosis, Tolerance Biomarkers, and Mechanisms in Microneedle Immunotherapy
Status: Not yet recruiting | Type: Observational
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Other Study IDs: PI24/00132; PI24/00132 (Other: Carlos III Health Institute)
Record Dates: First submitted 2025-05-13; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Food Allergies
Keywords: Vegetable food allergy; Allergy desensitization; Lipid Transfer Proteins
MeSH Terms: conditions — Food Hypersensitivity | interventions — Diet Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1. Patients on a maximum tolerated dose (MTD) diet.: To evaluate MTD, DBPCFC will be done with peach with skin and/or peach juice as described. The patient will remain under observation for at least 2 hours.
  Interventions: Procedure: Double-blind placebo-controlled oral challenge test (DBPCFC)
- Group 2. Allergic patients with dietary peach restriction.: Patients will take for one year, MTD of fresh peach or peach juice with a frequency of 3 times/week.
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Procedure: Double-blind placebo-controlled oral challenge test (DBPCFC) — Group 1. To evaluate MTD, DBPCFC will be done with peach with skin and/or peach juice as described. The patient will remain under observation for at least 2 hours.
  Groups: Group 1. Patients on a maximum tolerated dose (MTD) diet.
Other: Dietary intervention — Group 2. Patients will take for one year, MTD of fresh peach or peach juice with a frequency of 3 times/week.
  Groups: Group 2. Allergic patients with dietary peach restriction.

SUMMARY:
In relation to the prognosis of vegetable FA (VFA), in contrast to other food allergies (FA), which disappear naturally with time, VFA tends to persist into adulthood and to the appearance of new sensitizations to other vegetables. The paradigm of early intervention in patients with risk factors for developing FA has changed in recent years, with evidence that maintaining a controlled diet with foods with potential allergic risk in a population of children at risk has shown efficacy in early intervention. An important aspect would be the selection of the dose of the food to be included in the diet. In this sense, recent studies on the standardization of the double-blind placebo-controlled oral challenge test (DBPCFC) in allergic patients to Lipid Transfer Proteins (LTP) with known amounts of Pru p 3 (peach LTP), have observed that the maximum tolerated dose (MTD) was equivalent to 40 grams of peach with skin. Based on these results and those obtained in the pediatric population, this study aims to evaluate whether the maintenance in the diet of a DMT evaluated in a DBPCFC could influence tolerance (desensitization) to the food at both clinical and immunological levels.

ELIGIBILITY:
Inclusion Criteria:

* Women and men
* 14-65 years-old
* Peach allergy due to sensitization to LTP confirmed by skin tests and/or IgEe positive to Pru p 3.
* Sign informed consent.

Exclusion Criteria:

* Pregnant of lactating women.
* Patients with immunological diseases, mental illness or severe atopic dermatitis.
* Patients treated with immunomodulators and/or β-blockers
* Patients with forced expiratory volume (FEV1)<70%.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women and men aged 14-65 years with peach allergy due to sensitization to LTP confirmed by skin tests and/or IgEe positive to Pru p 3.
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Changes in the distribution of immune cell populations after MTD exposure | 1 year
  Study of the clinical and immunological implications of maintaining in the diet the maximum tolerated dose identified in a controlled food exposure test according to the sensitization profile to LTPs (Real-time pilot study).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Regional Universitario de Málaga, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No